CLINICAL TRIAL: NCT06505343
Title: Investigation of the Effect of Freezing Phenomenon on Gait Parameters and Pedobarographic Pressure Distribution in Patients With Parkinson's Disease
Brief Title: Effect of Freezing Phenomenon in Patients With Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Suleyman Korkusuz, Principal Investigator, Hacettepe University
Other Study IDs: e2d1895a2fd54888
Record Dates: First submitted 2024-05-06; First posted 2024-07-17 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Patients With Parkinson's Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Parkinson's patients with freezing phenomenon: Parkinson's patients with freezing phenomenon
- Parkinson's patients without freezing phenomenon: Parkinson's patients without freezing phenomenon
- Healthy: Healthy

SUMMARY:
Although the literature review indicates that plantar pressure may be related to freezing, there are not enough studies examining the effect of freezing phenomenon on pedobarographic pressure distribution and gait parameters. Therefore, the aim of our study is to examine the effect of freezing phenomenon on gait parameters and pedobarographic pressure distribution in patients with Parkinson's Disease.

DETAILED DESCRIPTION:
Individuals diagnosed with Idiopathic Parkinson's disease by a physician and healthy individuals with similar demographic characteristics will be included in the study. Individuals will be examined in 3 groups: a group of patients with Parkinson's Disease with freezing phenomenon, a group of patients with Parkinson's Disease without freezing phenomenon, and a healthy control group.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being between stage 2-3 according to the Modified Hoehn-Yahr Staging Scale
* Having a score of 24 or above from the Standardized Mini Mental Test

Exclusion Criteria:

* Presence of an additional neurological or psychiatric disease other than Parkinson's disease
* Presence of uncontrollable dyskinesia or motor fluctuations
* Presence of postural hypotension, vision problems (that cannot be compensated with the correct lens) or vestibular disorders that may affect balance
* Presence of cardiopulmonary diseases that may affect walking
* Presence of orthopedic problems and inflammatory arthritis (such as fractures, osteoporosis, osteomyelitis) that may cause limitation of movement and affect gait and evaluations

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Computerized Gait Evaluation System | Baseline
  This system allows the measurement of spatiotemporal features of gait.
Pressure distribution measurement platform | Baseline
  This system allows the measurement of dynamic foot pressure distribution with the pressure distribution measurement platform integrated into the system
Kinematic analysis | Baseline
  Kinematic analysis of the gait can be performed with the camera support within the system.
The freezing of gait questionnaire | Baseline
  This scale is a scale that evaluates freezing. This scale is related to patients' experiences, especially in the last week. One article describes the frequency of freezing seen in patients.

CONTACTS AND LOCATIONS:
Overall Officials: Süleyman Korkusuz, PhD, Principal Investigator — Atılım University; Büşra Seçkinoğulları Korkusuz, MSc, Study Chair — Ankara University; Ayşenur Özcan, Study Chair — Çankırı Karatekin University; Emine Nur Demircan, Msc, Study Chair — Hacettepe University; Ferdi Yavuz, Assoc.Prof, Study Chair — European University of Lefke; Bülent Elibol, Prof.Dr., Study Chair — Hacettepe University; Gül Yalçın Çakmaklı, Assoc.Prof, Study Chair — Hacettepe University; Ayla Fil Balkan, Assoc.Prof, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morris ME, Iansek R, Matyas TA, Summers JJ. The pathogenesis of gait hypokinesia in Parkinson's disease. Brain. 1994 Oct;117 ( Pt 5):1169-81. doi: 10.1093/brain/117.5.1169. PMID 7953597
- [Background] Giladi N, Nieuwboer A. Understanding and treating freezing of gait in parkinsonism, proposed working definition, and setting the stage. Mov Disord. 2008;23 Suppl 2:S423-5. doi: 10.1002/mds.21927. No abstract available. PMID 18668629